CLINICAL TRIAL: NCT01087086
Title: Reduction of the Metabolic Syndrome in Navarra-Spain (RESMENA-S) Through an Innovative Multidisciplinary Strategy Based on the Crononutrition and Dietary Training Concepts, in Addition to Both Dietary and Psychological Control
Brief Title: Reduction of the Metabolic Syndrome in Navarra-Spain
Acronym: RESMENA-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Hospital of Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESMENA-S
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2011-11

CONDITIONS: Metabolic Syndrome; Obesity; Diabetes; Cardiovascular Disease
Keywords: Metabolic syndrome; Oxidative stress; Proinflammatory state; Insulin resistance; Hypertension; Dyslipidemia; Mediterranean diet; Glycemic index; Hypocaloric diet; Hyperproteic diet; Macronutrient distribution; Antioxidant capacity of the diet; Crononutrition; Dietary and psychological support; Waist circumference
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Diabetes Mellitus; Cardiovascular Diseases; Insulin Resistance; Hypertension; Dyslipidemias | interventions — ANAPC16 protein, human; Adiposity; Heart Disease Risk Factors; American Heart Association

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crononutrition (Experimental): Dietary pattern:
  * Personalized diet
  * Caloric restriction (-30% Total energy intake)
  * High adherence to the Mediterranean Diet
  * Macronutrient distribution (30% Protein, 40% Carbohydrates and 30% Fat)
  * Low glycemic index/load
  * Increased antioxidant capacity of the diet
  Interventions: Behavioral: Crononutrition
- American Heart Association (Placebo Comparator): Dietary pattern:
  * Personalized diet
  * Caloric diet (-30% Total energy intake)
  * Macronutrients distribution according to the American Heart Association (AHA) guidelines
  Interventions: Behavioral: American Heart Association

INTERVENTIONS:
Behavioral: Crononutrition — After the recruitment and selection of the study participants, the study will consists of a 2-month nutritional intervention (Crononutrition versus AHA) followed by second 6-month period ("autonomy phase") in which the subjects of the study will continue with their ruled dietary patterns, but without any dietary or psychological support.
  Other Names: RYTHMONUTRITION; METABOLIC SYNDROME; OBESITY; DIABETES; CARDIOVASCULAR DISEASE; RESMENA-S
  Arms: Crononutrition
Behavioral: American Heart Association — After the recruitment and selection of the study participants, the study will consists of a 2-month nutritional intervention (Crononutrition versus AHA) followed by second 6-month period ("autonomy phase") in which the subjects of the study will continue with their ruled dietary patterns, but without any dietary or psychological support.
  Other Names: RESMENA-A
  Arms: American Heart Association

SUMMARY:
The purpose of this study is to determine whether a dietary pattern based on crononutrition and dietary training, together with dietary and psychological control, can reduce the body weight, improve the oxidative and inflammatory state in subjects with diagnosed metabolic syndrome features and can reduce the prevalence of the Metabolic syndrome in the population.

DETAILED DESCRIPTION:
The dietary pattern that characterizes the present nutritional intervention study is based on personalized diet, by elaborating tailoring-diets for each subject regarding his energetic needs and assuring a high adherence to the Mediterranean Diet. Moreover, the diet to be performed will be a hyperproteic diet to guarantee a satiety effect and a lower recovery of the lost weight, in accordance with the results derived from the main European study about nutrition (DIOGENES). The glycemic index/load will be also controlled in the study diet. The increase of the antioxidant capacity of the diet will be increased by the intake of fruits, walnuts and virgin olive oil among other antioxidant containing foods.

The present initiative, based on the traditional diet, aims to integrate the main results obtained from diverse observational epidemiological studies and interventional studies in the dietary pattern of the present study. At the same time, the study will apply the concept of crononutrition by selecting and distributing the foods thorough the day according the physiological needs of each individual.

In addition to the quantitative and qualitative composition of the diet, the study will take into account other important factors such as the behavior habits regarding the food, the frequency of consumption, the size of the eating portions, the distribution of the portions along the day, the feeling of fullness, the eating speed and so on. The aforementioned factors have recently been shown to be related to the gain of weight.

Other non dietary factors, such as smoking habits, sedentary life, socio-economic level, will be also controlled in the present study. Moreover, the project will integrate the dietary support together with psychological support due to the fact that the state of mind has been shown to be associated with the MS in some scientific publications.

ELIGIBILITY:
Inclusion Criteria:

* 35-70 years old
* Both sexes: Male and Female
* Metabolic Syndrome according to the IDF(2005)criteria:

Waist circumference cutoffs (male ≥94 cm or female ≥80 cm) plus any two of the following four factors:

1. Fasting glucose ≥5.55 mmol/L or use of antidiabetic medication
2. Systolic BP ≥130 mm Hg, diastolic BP ≥85 mm Hg, or use of antihypertensive medication
3. Fasting triglycerides ≥1.7 mm/L; and HDL-C <1.0 mm/L in men and <1.3 mm/L in women or specific treatment for this lipid abnormality

Exclusion Criteria:

* Recent follow-up of diets designed for weight loss
* Unstable weight in the past 3 months
* Alcoholic and drug dependence
* Hormonal treatment
* No stable pharmacological treatment
* Eating-disordered behaviors
* Severe physical or mental disability
* Pregnancy
* Terminal disease
* Institutionalization

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Body fat | One year
  Through this specific nutritional intervention program we will try to reduce the metabolic syndrome features such as waist circumference, body weight and adiposity.
  To evaluate the body composition, bioimpedance, DEXA and anthropometry methodology will be used at the beginning and after two months of intervention.
Lipid profile | One year
  To evaluate lipid improvements the following measurements will be taking into account:
  * Free fatty acids
  * Total cholesterol
  * HDL-cholesterol
  * LDL-cholesterol
Glucose Profile | One year
  To evaluate glucose improvements the following measurements will be taking into account:
  * Glucose
  * Insulin
  * HOMA

SECONDARY OUTCOMES:
Inflammation state | One year
  As secondary outcome some inflammatory markers will be analyzed:
  * CRP
  * IL-6
  * TNF-alpha
  * IL-18
  * PAI-1
  * Homocystein
Oxidative stress | One year
  As secondary outcome some oxidative stress markers will be analyzed:
  * MDA
  * LDL-OX
  * Total antioxidant capacity (TAC)
Psychological tests | January 2010-November 2011
  * Beck Depression Inventory
  * Stai Trait Anxiety Inventory
  * Mood thermometer visual analogue scale
  * Anxiety thermometer visual analogue scale
  * NEO personality inventory-revised test
Peripheral neurotransmitters | March-April 2013
  * Dopamine
  * Dopac
  * Serotonin
  * 5-Hydroxyindoleacetic acid
  * Noradrenaline
Epigenetics | April 2012-July 2014
  * DNA methylation
  * microRNAs expression
Fatty Liver biomarkers / Non invasive liver scoring system. | May 2016- January 2017
  Measurements in fatty liver biomarkers:
  Serum transaminases (AST & ALT (U/L)), GGT (U/L) and CK18 (U/L) concentrations will be measured in a fasting state at the beginning, at 2 months and at the end of the intervention.
  - A specificif Fatty Liver Index was calculated at the begining, at 2 months and at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: María Ángeles MA Zulet, PhD, Principal Investigator — University of Navarra; José Alfredo JA Martínez, PhD, RN, Study Director — University of Navarra; Itziar I Abete, PhD, Study Chair — University of Navarra; Lluis L Forga, PhD, Study Chair — Hospital of Navarra; Blanca Esther BE Martínez de Morentin, MD, Study Chair — University of Navarra; Santiago S Navas-Carretero, PhD, Study Chair — University of Navarra; Rocío R de la Iglesia, M.Sc, Study Chair — University of Navarra; Patricia P López Legarrea, M.Sc, Study Chair — University of Navarra; Isabel I Bondia-Pons, PhD, Study Chair — University of Navarra; Aurora A Perez Cornago, M.Sc, Study Chair — University of Navarra; José Luiz JL Marques-Rocha, M.Sc, Study Chair — Universidade Federal de Viçosa; Marcos M García-Lacarte, M.Sc, Study Chair — University of Navarra; Irene I Cantero, M.Sc, Study Chair — University of Navarra
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Hermsdorff HH, Zulet MA, Abete I, Martinez JA. Discriminated benefits of a Mediterranean dietary pattern within a hypocaloric diet program on plasma RBP4 concentrations and other inflammatory markers in obese subjects. Endocrine. 2009 Dec;36(3):445-51. doi: 10.1007/s12020-009-9248-1. PMID 19816812
- [Background] Puchau B, Zulet MA, de Echavarri AG, Hermsdorff HH, Martinez JA. Dietary total antioxidant capacity is negatively associated with some metabolic syndrome features in healthy young adults. Nutrition. 2010 May;26(5):534-41. doi: 10.1016/j.nut.2009.06.017. Epub 2009 Sep 26. PMID 19783122
- [Background] Perez-Matute P, Zulet MA, Martinez JA. Reactive species and diabetes: counteracting oxidative stress to improve health. Curr Opin Pharmacol. 2009 Dec;9(6):771-9. doi: 10.1016/j.coph.2009.08.005. Epub 2009 Sep 18. PMID 19766058
- [Background] Toledo E, de A Carmona-Torre F, Alonso A, Puchau B, Zulet MA, Martinez JA, Martinez-Gonzalez MA. Hypothesis-oriented food patterns and incidence of hypertension: 6-year follow-up of the SUN (Seguimiento Universidad de Navarra) prospective cohort. Public Health Nutr. 2010 Mar;13(3):338-49. doi: 10.1017/S1368980009991066. Epub 2009 Aug 6. PMID 19656442
- [Background] Sotos-Prieto M, Zulet MA, Corella D. [Scientific evidence of the mediterranean diet effects in determining intermediate and final cardiovascular disease phenotypes]. Med Clin (Barc). 2010 Jan 23;134(1):22-9. doi: 10.1016/j.medcli.2009.01.033. Epub 2009 May 19. Spanish. PMID 19457510
- [Background] Puchau B, Zulet MA, Gonzalez de Echavarri A, Navarro-Blasco I, Martinez JA. Selenium intake reduces serum C3, an early marker of metabolic syndrome manifestations, in healthy young adults. Eur J Clin Nutr. 2009 Jul;63(7):858-64. doi: 10.1038/ejcn.2008.48. Epub 2008 Nov 5. PMID 18985060
- [Background] Zulet MA, Puchau B, Navarro C, Marti A, Martinez JA. [Inflammatory biomarkers: the link between obesity and associated pathologies]. Nutr Hosp. 2007 Sep-Oct;22(5):511-27. Spanish. PMID 17970534
- [Background] Abete I, Parra MD, Zulet MA, Martinez JA. Different dietary strategies for weight loss in obesity: role of energy and macronutrient content. Nutr Res Rev. 2006 Jun;19(1):5-17. doi: 10.1079/NRR2006112. PMID 19079872
- [Background] Martinez MA, Puig JG, Mora M, Aragon R, O'Dogherty P, Anton JL, Sanchez-Villares T, Rubio JM, Rosado J, Torres R, Marcos J, Pallardo LF, Banegas JR; MAPA (Monitorizacion Ambulatoria de la Presion Arterial) Working Group. Metabolic syndrome: prevalence, associated factors, and C-reactive protein: the MADRIC (MADrid RIesgo Cardiovascular) Study. Metabolism. 2008 Sep;57(9):1232-40. doi: 10.1016/j.metabol.2008.04.017. PMID 18702949
- [Background] Sanchez-Chaparro MA, Calvo-Bonacho E, Gonzalez-Quintela A, Fernandez-Labandera C, Cabrera M, Sainz JC, Fernandez-Meseguer A, Banegas JR, Ruilope LM, Valdivielso P, Roman-Garcia J; Ibermutuamur Cardiovascular Risk Assessment (ICARIA) Study Group. Occupation-related differences in the prevalence of metabolic syndrome. Diabetes Care. 2008 Sep;31(9):1884-5. doi: 10.2337/dc08-0431. Epub 2008 Jun 20. PMID 18753667
- [Background] Babio N, Bullo M, Basora J, Martinez-Gonzalez MA, Fernandez-Ballart J, Marquez-Sandoval F, Molina C, Salas-Salvado J; Nureta-PREDIMED Investigators. Adherence to the Mediterranean diet and risk of metabolic syndrome and its components. Nutr Metab Cardiovasc Dis. 2009 Oct;19(8):563-70. doi: 10.1016/j.numecd.2008.10.007. Epub 2009 Jan 26. PMID 19176282
- [Background] Abete I, Parra D, Martinez JA. Legume-, fish-, or high-protein-based hypocaloric diets: effects on weight loss and mitochondrial oxidation in obese men. J Med Food. 2009 Feb;12(1):100-8. doi: 10.1089/jmf.2007.0700. PMID 19298202
- [Background] Goyenechea E, Parra D, Crujeiras AB, Abete I, Martinez JA. A nutrigenomic inflammation-related PBMC-based approach to predict the weight-loss regain in obese subjects. Ann Nutr Metab. 2009;54(1):43-51. doi: 10.1159/000205319. Epub 2009 Feb 27. PMID 19246894
- [Background] Abete I, Parra D, Martinez JA. Energy-restricted diets based on a distinct food selection affecting the glycemic index induce different weight loss and oxidative response. Clin Nutr. 2008 Aug;27(4):545-51. doi: 10.1016/j.clnu.2008.01.005. Epub 2008 Mar 4. PMID 18308431
- [Derived] Cantero I, Abete I, Del Bas JM, Caimari A, Arola L, Zulet MA, Martinez JA. Changes in lysophospholipids and liver status after weight loss: the RESMENA study. Nutr Metab (Lond). 2018 Jul 17;15:51. doi: 10.1186/s12986-018-0288-5. eCollection 2018. PMID 30026784
- [Derived] de la Iglesia R, Mansego ML, Sanchez-Muniz FJ, Zulet MA, Martinez JA. Arylesterase activity is associated with antioxidant intake and paraoxonase-1 (PON1) gene methylation in metabolic syndrome patients following an energy restricted diet. EXCLI J. 2014 Apr 9;13:416-26. eCollection 2014. PMID 26417268
- [Derived] Garcia-Lacarte M, Milagro FI, Zulet MA, Martinez JA, Mansego ML. LINE-1 methylation levels, a biomarker of weight loss in obese subjects, are influenced by dietary antioxidant capacity. Redox Rep. 2016 Mar;21(2):67-74. doi: 10.1179/1351000215Y.0000000029. Epub 2016 Feb 15. PMID 26197243
- [Derived] Bondia-Pons I, Martinez JA, de la Iglesia R, Lopez-Legarrea P, Poutanen K, Hanhineva K, Zulet Mde L. Effects of short- and long-term Mediterranean-based dietary treatment on plasma LC-QTOF/MS metabolic profiling of subjects with metabolic syndrome features: The Metabolic Syndrome Reduction in Navarra (RESMENA) randomized controlled trial. Mol Nutr Food Res. 2015 Apr;59(4):711-28. doi: 10.1002/mnfr.201400309. Epub 2015 Feb 5. PMID 25641909
- [Derived] Perez-Cornago A, de la Iglesia R, Lopez-Legarrea P, Abete I, Navas-Carretero S, Lacunza CI, Lahortiga F, Martinez-Gonzalez MA, Martinez JA, Zulet MA. A decline in inflammation is associated with less depressive symptoms after a dietary intervention in metabolic syndrome patients: a longitudinal study. Nutr J. 2014 Apr 24;13:36. doi: 10.1186/1475-2891-13-36. PMID 24762259
- [Derived] Lopez-Legarrea P, de la Iglesia R, Crujeiras AB, Pardo M, Casanueva FF, Zulet MA, Martinez JA. Higher baseline irisin concentrations are associated with greater reductions in glycemia and insulinemia after weight loss in obese subjects. Nutr Diabetes. 2014 Feb 24;4(2):e110. doi: 10.1038/nutd.2014.7. PMID 24567125
- [Derived] Perez-Cornago A, Lopez-Legarrea P, de la Iglesia R, Lahortiga F, Martinez JA, Zulet MA. Longitudinal relationship of diet and oxidative stress with depressive symptoms in patients with metabolic syndrome after following a weight loss treatment: the RESMENA project. Clin Nutr. 2014 Dec;33(6):1061-7. doi: 10.1016/j.clnu.2013.11.011. Epub 2013 Nov 22. PMID 24314875
- [Derived] Lopez-Legarrea P, Mansego ML, Zulet MA, Martinez JA. SERPINE1, PAI-1 protein coding gene, methylation levels and epigenetic relationships with adiposity changes in obese subjects with metabolic syndrome features under dietary restriction. J Clin Biochem Nutr. 2013 Nov;53(3):139-44. doi: 10.3164/jcbn.13-54. Epub 2013 Oct 31. PMID 24249967
- [Derived] Lopez-Legarrea P, de la Iglesia R, Abete I, Bondia-Pons I, Navas-Carretero S, Forga L, Martinez JA, Zulet MA. Short-term role of the dietary total antioxidant capacity in two hypocaloric regimes on obese with metabolic syndrome symptoms: the RESMENA randomized controlled trial. Nutr Metab (Lond). 2013 Feb 13;10(1):22. doi: 10.1186/1743-7075-10-22. PMID 23406163
- [Derived] Zulet MA, Bondia-Pons I, Abete I, de la Iglesia R, Lopez-Legarrea P, Forga L, Navas-Carretero S, Martinez JA. The reduction of the metabolyc syndrome in Navarra-Spain (RESMENA-S) study: a multidisciplinary strategy based on chrononutrition and nutritional education, together with dietetic and psychological control. Nutr Hosp. 2011 Jan-Feb;26(1):16-26. PMID 21519726